CLINICAL TRIAL: NCT00863161
Title: A Phase I, Open Label, Non-randomized, Parallel Group, Pharmacokinetic Study in Subjects With Normal Renal Function, Moderate or Severe Renal Impairment Receiving a Single Dose of Oral 130 mg AZD3355
Brief Title: Renal Impairment Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Debra G. Silberg, MD, PhD, Medical Science Director, AZD3355, AstraZeneca Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D9120C00022; EudraCTnr 2008-007471-25
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Reflux; Renal Excretion
Keywords: Safety; tolerability; exposure; healthy; renally impaired subjects
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — lesogaberan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): AZD3355 65 + 65 mg capsule
  Interventions: Drug: AZD3355

INTERVENTIONS:
Drug: AZD3355 — capsule, oral, single dose
  Other Names: Lesogaberan

SUMMARY:
The purpose of this study is to see how quickly AZD3355 is taken up in to the blood and leaves the blood in people with normal kidney function or with different degrees of reduced kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent
* Subjects should have either normal renal function or have a moderate renal impairment or severe renal impairment

Exclusion Criteria:

* History of heart disease
* Unstable or clinically significant other disorders such as respiratory, hepatic, metabolic, psychiatric or gastrointestinal disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic blood samples | 15 samples during 0-72 hours

SECONDARY OUTCOMES:
Pharmacokinetic urine samples | 8 samples during 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Kuhn, MD, Principal Investigator — Quintiles AB, Phase I Services, Strandbodgatan 1, 753 23 Uppsala, Sweden
Locations (3):
- Sweden (3):
  - Research Site, Linköping
  - Research Site, Luleå
  - Research, Uppsala